CLINICAL TRIAL: NCT04805723
Title: Comparison of Video-Assisted Thoracoscopy Surgery and Thoracotomy on Cardiorespiratory Parameters in Patients With Pulmonary Nodules
Brief Title: Effects of Surgery Types in Patients With Pulmonary Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof.Dr, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Gazi University 509
Record Dates: First submitted 2021-02-28; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary Nodule
Keywords: pulmonary nodule; pulmonary function; functional exercise capacity; physical activity; respiratory muscle strength; respiratory muscle endurance; quality of life
MeSH Terms: conditions — Motor Activity | interventions — Thoracic Surgery, Video-Assisted; Thoracotomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with pulmonary nodule scheduled VATS (Experimental): Patients with pulmonary nodule scheduled VATS were included in this study. Inclusion and exclusion criteria were considered.
  Pulmonary function (spirometry), functional exercise capacity (6-minute walk test (6-MWT); 6-minute stepper test (6-MST)), physical activity level (metabolic holter), respiratory (maximal inspiratory and expiratory pressures (MIP-MEP); mouth pressure device) and peripheral muscle strength (dynamometer), inspiratory muscle endurance (incremental loading test), quality of life (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTCQOL)), fatigue (Fatigue Severity Scale), dyspnea perception (Modified Medical Research Council dyspnea scale (MMRC)) and pain severity (Visual Analog Scale) were assessed before VATS and average two weeks after surgery.
  Interventions: Procedure: VATS
- Patients with pulmonary nodule scheduled thoracotomy (Experimental): Patients with pulmonary nodule scheduled thoracotomy were included in this study. Inclusion and exclusion criteria were considered.
  Pulmonary function (spirometry), functional exercise capacity (6-minute walk test (6-MWT); 6-minute stepper test (6-MST)), physical activity level (metabolic holter), respiratory (maximal inspiratory and expiratory pressures (MIP-MEP); mouth pressure device) and peripheral muscle strength (dynamometer), inspiratory muscle endurance (incremental loading test), quality of life (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTCQOL)), fatigue (Fatigue Severity Scale), dyspnea perception (Modified Medical Research Council dyspnea scale (MMRC)) and pain severity (Visual Analog Scale) were assessed before VATS and average two weeks after surgery.
  Interventions: Procedure: Thoracotomy

INTERVENTIONS:
Procedure: VATS — Video-assisted thoracoscopic surgery is a minimal invasive technique in which used to diagnose or treat for lung diseases. During this surgery, one or two small incisions are opened via camera and surgical instruments in patient's chest wall. Thus, less muscle and nerve tissue are damaged.
  Thoracotomy is an open surgical technique in which allowing visualization of the inside of the thorax. During this surgery, an incision in patient's chest wall is made between the ribs and some muscles important for respiration are cutted to remove a part of lung.
  Arms: Patients with pulmonary nodule scheduled VATS
Procedure: Thoracotomy — Thoracotomy is an open surgical technique in which allowing visualization of the inside of the thorax. During this surgery, an incision in patient's chest wall is made between the ribs and some muscles important for respiration are cutted to remove a part of lung.
  Arms: Patients with pulmonary nodule scheduled thoracotomy

SUMMARY:
The investigators aimed to compare the pre-post operative effects of video-assisted thoracoscopy surgery (VATS) and thoracotomy on pulmonary function, exercise capacity, physical activity level, respiratory and peripheral muscle strength, inspiratory muscle endurance, quality of life, fatigue, dyspnea perception and pain in patients with pulmonary nodules.

DETAILED DESCRIPTION:
According to global cancer statistics, lung cancer accounts for 11.6% of all cancer cases and it is the most common type of cancer in the world. Surgery is the primary treatment approach, especially in early stages lung cancer. Cardiopulmonary fitness of patients with lung cancer is lower than healthy individuals due to the disease itself and treatments. Pulmonary function, exercise capacity and physical activity level are affected in lung cancer depending on the resected lung tissue and the type of surgery. VATS and thoracotomy surgeries, which are the most preferred techniques in lung cancer, have advantages and disadvantages over each other. There are few studies compared the early effects of two surgeries on the pulmonary function, exercise capacity, physical activity, quality of life and fatigue. And also, no study compared the effects of two surgeries on respiratory muscle endurance and peripheral muscle strength, previously.

According to sample size calculation, at least 15 patients with pulmonary lesion both VATS and thoracotomy groups would be included in the study. The demographic, physical and physiological characteristics were recorded from the patient files. Pulmonary function, functional exercise capacity, physical activity level, respiratory and peripheral muscle strength, inspiratory muscle endurance, quality of life, fatigue, dyspnea perception and pain were evaluated pre and two weeks after postoperative term. Primary outcomes were pulmonary function, functional exercise capacity and physical activity level. Secondary outcomes were respiratory and peripheral muscle strength, inspiratory muscle endurance, quality of life, fatigue, dyspnea perception and pain.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-80 years of age,
* Patients with pulmonary nodule who were planned lobectomy surgery with one of VATS or thoracotomy techniques,
* Being able to walk,

Exclusion Criteria:

* Any type of surgery planned except lobectomy,
* Having heart failure or atrial fibrillation,
* Having acute viral infections during all assessment,
* History of acute myocard infarction within last six months,
* Uncontrolled diabetes or hypertension,
* Having orthopedic, neurological and psychological disorders that influence the results of study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test (Forced expiratory volume in one second) | first day
  Forced expiratory volume in one second was evaluated with spirometry according American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. The value was represented as percentages.
Pulmonary function test (Forced vital capacity) | first day
  Forced vital capacity was evaluated with spirometry according to ATS and ERS criteria. The value was represented as percentages.
Pulmonary function test (Forced expiratory volume in one second/Forced vital capacity) | first day
  Forced expiratory volume in one second/Forced vital capacity was evaluated with spirometry according to ATS and ERS criteria. The value was represented as percentages.
Pulmonary function test (Peak expiratory flow) | first day
  Peak expiratory flow was evaluated with spirometry according to ATS and ERS criteria. The value was represented as percentages.
Pulmonary function test (Flow rate 25-75% of forced expiratory volume) | first day
  Flow rate 25-75% of forced expiratory volume was evaluated with spirometry according to ATS and ERS criteria. The value was represented as percentages.
6-minute walk test | first day
  6-minute walk test were used to assess functional exercise capacity according to the guidelines. The test was repeated twice in the same day with 30 min interval. The highest distance was recorded for analysis.
6-minute stepper test | second day
  6-minute stepper test were used to assess functional exercise capacity according to the guidelines. The height of the stepper used for test was 20 cm. A cycle of up and down was define as one step. The number of steps was recorded for analysis.
Physical activity assessment | second day
  Total energy expenditure (joules/day), active energy expenditure (>3.0 metabolic equivalents (METs)) (joules/day), physical activity duration (>3.0 METs) (min/day), average MET (METs/day), number of steps (steps/day), lying down (min/day) and sleeping duration (min/day) were measured to interpret the physical activity level of the patients via metabolic holter device. The metabolic holter was worn over triceps brachii muscle of non-dominant extremity for two consecutive days. The patients' activity level were categorized according to number of steps and average MET sums.

SECONDARY OUTCOMES:
Inspiratory muscle strength test | first day
  Maximal inspiratory pressure (MIP) was performed to evaluate respiratory muscle strength. Evaluation was done by using portable mouth pressure device accordance with the guidelines. The MIP was measured at residual volume after maximal expiration. The measurements were repeated at least seven times for technically acceptable value.
Expiratory muscle strength test | first day
  Maximal expiratory pressure (MEP) was performed to evaluate respiratory muscle strength. Evaluation was done by using portable mouth pressure device accordance with the guidelines. The MEP was measured from total lung capacity after maximal inspiration. The measurements were repeated at least seven times for technically acceptable value.
Peripheral muscle strength test | first day
  Shoulder abduction, shoulder flexion, elbow extension, quadriceps femoris muscle strength and hand grip strength were evaluated using a hand held dynamometer. The measurements of each muscle were repeated bilaterally three times.
Inspiratory muscle endurance test | second day
  Inspiratory muscle endurance test were performed using respiratory muscle trainer (POWERbreathe) according to incremental threshold loading test protocol. The endurance test was started at thirty percentage of MIP and each two minutes the load of test was increased by ten percentage of MIP. The highest percentage of MIP could be reached and sustained for at least 1 min was defined as maximal load and time were recorded for analysis.
Modified borg scale | first and second day
  This scale was used to evaluate dyspnea and fatigue perception during 6-minute walk test and 6-minute stepper test. It was scored between 0 and 10. The lowest value was 0 which was meant no dyspnea or fatigue and the highest value was 10 which was meant worse and severe dyspnea and fatigue.
Quality of life scale | first day
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 version3.0 (Turkish version of scale) were used. The questionnaire comprise of 30 items in which five scales and several single items are graded from 1 (not at all) to 4 (very much) except for 29-30 items. All scales and items' scores are expressed by transforming to a 0-100 scale. Higher values except symptom scale represent higher quality of life. The minimum value was '0' and the maximum value was '100'. The highest value was meant better quality of life. The highest value for symptom scale was meant worse symptom.
Fatigue | second day
  Fatigue severity scale (Turkish version of scale) were applied. This one-dimensional scale compose of nine items scored between 1 (completely disagree) and 7 (completely agree). The minimum total value was 7 and the maximum total value was 63. The cut-off value for severe fatigue was 36 and the highest total value is meant severe fatigue.
Dyspnea perception | first day
  The Modified Medical Research Council dyspnea scale were performed to determine dyspnea perception during daily living activities. This categorical scale consisting of five expressions are scored from '0' to '4'. The minimum value was 0 which means no complain about dyspnea apart from strenuous exercise; the maximum value was 4 which means too breathless for leaving the house or dyspnea while getting dressed. The highest value was refered to severe shortness of breath during activities of daily living.
Pain severity | second day
  To evaluate pain severity, visual analog scale were used. The minimum value was 0 mm (no pain) and the maximum value was 100 mm (worst pain). The highest score was 100 mm which was meant worse pain severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ece BAYTOK, MsC., Study Chair — Gazi University; Zeliha ÇELİK, MsC., Principal Investigator — Gazi University; Merve ŞATIR TÜRK, MD., Principal Investigator — Gazi University; Ali ÇELİK, Assoc. Prof., Principal Investigator — Gazi University; İsmail Cüneyt KURUL, Prof. Dr., Principal Investigator — Gazi University; Meral Boşnak GÜÇLÜ, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Health Science, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Cavalheri V, Jenkins S, Cecins N, Gain K, Phillips M, Sanders LH, Hill K. Impairments after curative intent treatment for non-small cell lung cancer: a comparison with age and gender-matched healthy controls. Respir Med. 2015 Oct;109(10):1332-9. doi: 10.1016/j.rmed.2015.08.015. Epub 2015 Aug 29. PMID 26342839
- [Result] Nagamatsu Y, Maeshiro K, Kimura NY, Nishi T, Shima I, Yamana H, Shirouzu K. Long-term recovery of exercise capacity and pulmonary function after lobectomy. J Thorac Cardiovasc Surg. 2007 Nov;134(5):1273-8. doi: 10.1016/j.jtcvs.2007.06.025. PMID 17976462
- [Result] Kaseda S, Aoki T, Hangai N, Shimizu K. Better pulmonary function and prognosis with video-assisted thoracic surgery than with thoracotomy. Ann Thorac Surg. 2000 Nov;70(5):1644-6. doi: 10.1016/s0003-4975(00)01909-3. PMID 11093502
- [Result] Cheng X, Onaitis MW, D'amico TA, Chen H. Minimally Invasive Thoracic Surgery 3.0: Lessons Learned From the History of Lung Cancer Surgery. Ann Surg. 2018 Jan;267(1):37-38. doi: 10.1097/SLA.0000000000002405. No abstract available. PMID 28692471
- [Result] Upham TC, Onaitis MW. Video-assisted thoracoscopic surgery versus robot-assisted thoracoscopic surgery versus thoracotomy for early-stage lung cancer. J Thorac Cardiovasc Surg. 2018 Jul;156(1):365-368. doi: 10.1016/j.jtcvs.2018.02.064. Epub 2018 Mar 2. No abstract available. PMID 29921098
- [Result] Park TY, Park YS. Long-term respiratory function recovery in patients with stage I lung cancer receiving video-assisted thoracic surgery versus thoracotomy. J Thorac Dis. 2016 Jan;8(1):161-8. doi: 10.3978/j.issn.2072-1439.2016.01.14. PMID 26904225
- [Result] Granger CL, Parry SM, Edbrooke L, Denehy L. Deterioration in physical activity and function differs according to treatment type in non-small cell lung cancer - future directions for physiotherapy management. Physiotherapy. 2016 Sep;102(3):256-63. doi: 10.1016/j.physio.2015.10.007. Epub 2015 Oct 23. PMID 26597694
- [Result] Schwartz RM, Yip R, Flores RM, Olkin I, Taioli E, Henschke C; I-ELCAP Investigators. The impact of resection method and patient factors on quality of life among stage IA non-small cell lung cancer surgical patients. J Surg Oncol. 2017 Feb;115(2):173-180. doi: 10.1002/jso.24478. Epub 2016 Oct 28. PMID 27790715
- [Result] Nomori H, Kobayashi R, Fuyuno G, Morinaga S, Yashima H. Preoperative respiratory muscle training. Assessment in thoracic surgery patients with special reference to postoperative pulmonary complications. Chest. 1994 Jun;105(6):1782-8. doi: 10.1378/chest.105.6.1782. PMID 8205877